CLINICAL TRIAL: NCT06573580
Title: Pilot Project for the Primary Health Management of Chronic Obstructive Pulmonary Disease
Brief Title: Primary Health Management for Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, Deputy Director of the National Center for Respiratory Medicine, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-HX-59
Record Dates: First submitted 2024-07-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Disease; Chronic Obstructive Pulmonary Disease
Keywords: Primary Health Management; Health Economic Evaluation; Efficacy; Community-based
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual primary health care for COPD (No Intervention)
- The essential public health primary care for COPD (Experimental)
  Interventions: Other: The essential public health service（EPHS）for COPD

INTERVENTIONS:
Other: The essential public health service（EPHS）for COPD — Each group plans to recruit 3,000 participants. For the intervention group, the community-based management includes adding COPD management-related content to the primary public health service. This includes: Providing at least four follow-ups during the project at the 3rd, 6th, 9th, and 12th months. During each follow-up, patients must complete the "COPD Patient Follow-up Questionnaire" and receive oral health education and targeted clinical advice from the general practitioner (GP). In addition, the GPs must also distribute educational booklets and materials, record symptom assessment results and acute exacerbation situations, and provide targeted clinical advice and clinical decisions to the COPD patients according to the checklist of Chinese guideline for management of COPD in primary care. At the baseline and the last follow-up, patients need to undergo a routine physical examination, pulmonary function test, and bronchodilator test at their community health centers
  Arms: The essential public health primary care for COPD

SUMMARY:
The core objective of the "Pilot Project for the Primary Health Management of Chronic Obstructive Pulmonary Disease (COPD)" is to explore a primary health management model and service standards that are suitable for COPD patients and aligned with grassroots realities. It also aims to enhance the capability of primary healthcare institutions in the prevention and management of chronic respiratory diseases. The primary outcomes are to evaluate the efficacy and cost-effectiveness of COPD Essential Public Health Services (EPHS) intervention in communities in China.

Participants are already receiving intervention B, "Usual primary health care," as part of their regular medical care under the current health policy. Researchers will compare intervention A, which is"the EPHS for COPD", with intervention B to determine if intervention A performs better in COPD management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 35 years.
2. Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) according to the 2024 GOLD guidelines.
3. Post-bronchodilator FEV1(Forced Expiratory Volume in one second) predicted ≥ 30%.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Contraindications for pulmonary function tests, including:

   * Recent myocardial infarction, stroke, or shock within the past 3 months.
   * Severe heart failure, severe arrhythmias, or unstable angina within the past 4 weeks.
   * Recent major hemoptysis within the past 4 weeks.
   * Major thoracic, abdominal, or ophthalmic surgery within the past 3 months.
   * Psychiatric disorders requiring antipsychotic medication or with a history of seizures requiring medication.
   * Cognitive impairment, including dementia or severe comprehension deficits.
   * Uncontrolled hypertension (systolic blood pressure > 200 mmHg, diastolic blood pressure > 100 mmHg).
   * Resting heart rate > 120 beats per minute.
   * Presence of aortic aneurysm.
   * Severe hyperthyroidism.
   * Pregnancy or lactation.
   * Respiratory tract infections (e.g., tuberculosis, influenza, pneumonia) within the past month.
   * Presence of pneumothorax, large pulmonary bullae not scheduled for surgery, or tympanic membrane perforation.
3. Currently participating in, or planning to participate in, any other COPD health management or clinical intervention projects during the study period.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Acute exacerbation frequency | 12 months
  The number of exacerbations occurred
Self-rated Quality of Life | 12 months
  Quality of life measured by the EQ-5D-5L (EuroQol-5 Dimensions-5 Levels) questionnaire. It consists of two parts:
  Descriptive System: This includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels, ranging from no problems to extreme problems.
  Visual Analog Scale (VAS): This is a scale from 0 to 100, where 0 represents the worst possible health state and 100 represents the best possible health state.
  Scores from the descriptive system can be combined into a single health index value, while the VAS provides an immediate self-assessment of the respondent's health status. Higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Change in lung function | 6 months 12 months
  Decline in forced expiratory rate in one second (FEV1) before use of bronchodilator.
Degree of dyspnea (daily activity) | 12 months
  Measured by Modified Medical Research Council (mMRC) Dyspnea Questionnaire Minimum Value: 0 (no dyspnea) Maximum Value: 4 (severe dyspnea) It specifically assesses dyspnea based on the activity level at which shortness of breath occurs, ranging from 0 to 4. A score of 4 indicates that the patient experiences dyspnea with minimal activity, representing the most severe breathlessness.
Oxygen desaturation | 12 months
  SpO2 measured by a pulse oximeter.

OTHER OUTCOMES:
Nicotine dependence | 12 months
  Measured by Fagerström Test for Nicotine Dependence (FTND); Minimum Value: 0 (no dependence); Maximum Value: 10 (high dependence); The FTND is a widely used clinical tool to assess the level of nicotine dependence. It consists of 6 questions, each with answers assigned different point values. The cumulative score determines the level of nicotine dependence. Higher cumulative scores indicate greater nicotine dependence.
Healthcare expenditure for COPD | 12 months
  An online survey questionnaire to collect indirect and direct non-medical costs for COPD treatment, along with data obtained from the Chinese National Healthcare Security Administration (NHSA) for the direct costs of treating and managing COPD.
Clinic or emergency utilization | 6 months
  Clinic or emergency utilization in the past six months and clinic types were collected by an online survey questionnaire and from the Chinese National Healthcare Security Administration (NHSA).
Knowledge of Primary Health Care Providers | 12 months
  It is an online survey questionnaire designed by our team to explore the knowledge level of primary care physicians in China on COPD. The questionnaire includes components on COPD risk factors, screening, diagnosis, treatment and control, and public education.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, Principal Investigator — China-Japan Friendship Hospital; Chen Wang, Study Chair — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No